CLINICAL TRIAL: NCT03470415
Title: Relation of Epicardial Fat and Diabetic Nephropathy in Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Azeem Mohamed, Principle investigator, Assiut University
Other Study IDs: EPICARDIALNEPHRO
Record Dates: First submitted 2018-03-11; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Days

GROUPS / COHORTS (3):
- Group A: Patients with type 2 diabetes milletus with normoalbuminuria.
- Group B: Patients with type 2 diabetes milletus with microalbuminuria.
- Group C: Patients with type 2 diabetes milletus with macroalbuminuria.

SUMMARY:
The heart and vessels are surrounded by layers of adipose tissue, which is a complex organ composed of adipocytes, stromal cells, macrophages, and a neuronal network, all nourished by a rich microcirculation. The layers of adipose tissue surrounding the heart can be subdivided into intra- and extra-pericardial fat. Their thicknesses and volumes can be quantified by echocardiography and computed tomography or magnetic resonance imaging, respectively. The term extrapericardial fat defines thoracic adipose tissue external to the parietal pericardium. It originates from primitive thoracic mesenchymal cells and thus derives its blood supply from noncoronary sources. Intrapericardial fat is further subdivided into epicardial and pericardial fat. Anatomically, epicardial and pericardial adipose tissues are clearly different. Epicardial fat is located between the outer wall of the myocardium and the visceral layer of pericardium.

DETAILED DESCRIPTION:
The epicardial fat layer originates from mesothelial cells and hence obtains its vascular supply from the coronary arteries. Much of the importance within the epicardial fat is its anatomical closeness to the myocardium and the fact that the two tissues share the same microcirculation. Epicardial fat is a metabolically active organ that secrets numerous bioactive substances, which may alter cardiac function. This small, visceral fat depot had been accepted as a rich source of free fatty acids and a number of bioactive molecules, such as adiponectin, resistin and inflammatory cytokines, which could lead to the coronary endothelial dysfunction. Furthermore, epicardial adipose mass might reflect intra-abdominal visceral fat. Epicardial adipose tissue is also clinically related to left ventricular mass and other features of the metabolic syndrome, such as concentrations of LDL cholesterol, fasting insulin and adiponectin, and arterial blood pressure. Epicardial fat thickness can be visualized and measured with two-dimensional (2D) echocardiography. Standard parasternal long-axis and short-axis views from 2D images permit the most accurate measurement of epicardial fat thickness on the right ventricle, with optimal cursor beam orientation in each view. Echocardiographically, epicardial fat is generally identified as the relatively echo-free space between the outer wall of the myocardium and the visceral layer of pericardium; its thickness is measured perpendicularly on the free wall of the right ventricle at end-systole in 3 cardiac cycles. Because it is compressed during diastole, epicardial fat thickness is best measured at end-systole at the point on the free wall of the right ventricle at which the ultrasound beam is oriented in a perpendicular manner, using the aortic annulus as an anatomic landmark. Epicardial fat thickness can be also appear as hyperechoic space, if in large amount (>15 mm). Maximum epicardial fat thickness is measured from 2D parasternal long axis images at the point on the free wall of the right ventricle along the midline of the ultrasound beam, perpendicular to the aortic annulus, used as an anatomic landmark for this view. For midventricular parasternal short-axis assessment, maximum epicardial fat thickness is measured from 2D images on the right ventricular free wall along the midline of the ultrasound beam perpendicular to the interventricular septum at midchordal and tip of the papillary muscle level, as anatomic landmarks. The average value of 3 cardiac cycles from each echocardiographic view is determined. The majority of population based clinical studies have reported excellent interobserver and intraobserver agreement for epicardial fat thickness measurement. Echocardiographic epicardial fat measurement may have some advantages as an index of high cardiometabolic risk. It is a direct measure of visceral fat rather than an anthropometric measure, such as waist circumference, that includes muscle and skin layers. The echocardiographic measurement of epicardial fat provides a more sensitive and specific measure of true visceral fat content, avoiding the possible confounding effect of increased subcutaneous abdominal fat. It is an objective, noninvasive, readily available, and certainly less expensive measure of visceral fat than MRI or CT. Visceral cardiac fat can be quantified fairly precisely compared with ectopic fat deposition in organs such as the liver, which can be described only qualitatively unless expensive measurements are made, such as CT or MRI. Echocardiographic epicardial fat is a direct measure of ectopic fat deposition, whereas anthropometric measures can be associated only with ectopic fat deposition. It can be measured even from echocardiograms that were not specifically performed to optimize the measurement of epicardial fat. It can be quantified with other echocardiographic parameters, such left ventricular mass and ejection fraction, traditionally associated with cardiovascular risk. Echocardiographic epicardial fat could be a more reliable quantitative therapeutic marker during interventions modulating and reducing visceral adiposity. Diabetic nephropathy or diabetic kidney disease is a syndrome characterized by the presence of pathological quantities of urine albumin excretion, diabetic glomerular lesions, and loss of glomerular filtration rate (GFR) in diabetics. Incipient nephropathy is the initial presence of low but abnormal amounts of urine albumin, referred to as microalbuminuria (persistent albuminuria at level 30-299 mg/24 hours), while overt nephropathy or macroalbuminuria (persistent albuminuria at level 300 mg/24 hours).

ELIGIBILITY:
Inclusion Criteria:

All patients attends to internal medicine, cardiology or nephrology outpatient clinics with the following criteria:

1. Patients who are older than 30.
2. Patients who are younger than 65.
3. Patients with type 2 diabetes milletus.
4. Patients with renal complaints (loin pain, frequency, ….).
5. No sex predilection.

Exclusion Criteria:

1. Age:

   Patients who are less than 30 years or more than 65 years.
2. Patients with type 1 diabetes milletus or diabetes insipidus. 3. Patients with cardiac diseases: A. Patients with cardiac diseases ( coronary artery disease, heart failure, myocardial infarction, infection,…) or history of cardiac problem or previous intervention (PCI,..) will be excluded from our study.

B. Patients with cardiac congenital anomalies. 4. Patients with active infections. 5- Patients with autoimmune diseases: As rheumatoid arthritis or systemic lupus. 6- Patients with acute diabetic complications. 7- Patients with a family history of kidney failure. 8- Patients with other causes of nephropathy will be excluded as: A. Liver cirrhosis to exclude hepatorenal syndrome. B. Autoimmune diseases as lupus nephritis. C. History of excessive analgesics intake. D. End stage kidney disease (chronic renal failure on dialysis).

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All type 2 diabetic patients attends to internal medicine, cardiology or nephrology outpatient clinics
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of protein in urine | 1 day
  Urine analysis (for protein and creatinine): 24 hrs urine sample will be collected from all patients to detect presence and amount of protein in urine by dipstick or albumin in urine kits.
epicardial fat thickness measurement | 1 day
  Echocardiography: Two dimensional echocardiography perpendicularly on the free wall of the right ventricle at end-systole in 3 cardiac cycles will be performed to all patients to measure the epicardial fat thickness.

SECONDARY OUTCOMES:
laboratory tests | 7 days
  Fasting blood glucose, Blood sample for kidney function test, Blood sample for liver function test, C-reactive protein, complete blood count (blood sample on EDTA for calculating neutrophil lymphocyte ratio and platelet lymphocyte ratio) and HbA1c.
Imaging | 3 days
  Abdominal ultrasound to assess the kidney and other abdominal organs condition, CT for selected cases only and echocardiography to assess the heart and great vessels condition and detect any disease or abnormality.
Calculation of GFR | 1 day
  eGFR (Cockcroft-Gault equation) will be calculated by the following equation: GFR(ml/min)= ((140- age)Weight (kg))/(72XS.Cr (mg/dl)) For women,multiply with 0.85.
  *As weight in kilograms and creatinine in mg/dl. Patients will be instructed to fast overnight and not to eat cooked meat before the test.
Full history taking | 1 day
  Personal history: name, age, sex,…. and Disease history: onset, course, duration and stability, History of previous treatment and when it has been stopped and Family history of diabetes millets, cardiac or renal diseases will be taken
General examination | 1 day
  General clinical examination will be carried out to detect any associated abnormalities in other body systems.
Electrocardiogram | 1 day
  to assess the heart condition

REFERENCES:
- [Background] Meenakshi K, Rajendran M, Srikumar S, Chidambaram S. Epicardial fat thickness: A surrogate marker of coronary artery disease - Assessment by echocardiography. Indian Heart J. 2016 May-Jun;68(3):336-41. doi: 10.1016/j.ihj.2015.08.005. Epub 2016 Jan 18. PMID 27316487
- [Background] Iacobellis G, Willens HJ. Echocardiographic epicardial fat: a review of research and clinical applications. J Am Soc Echocardiogr. 2009 Dec;22(12):1311-9; quiz 1417-8. doi: 10.1016/j.echo.2009.10.013. PMID 19944955
- [Background] Lim AKh. Diabetic nephropathy - complications and treatment. Int J Nephrol Renovasc Dis. 2014 Oct 15;7:361-81. doi: 10.2147/IJNRD.S40172. eCollection 2014. PMID 25342915
- [Background] Akbas EM, Demirtas L, Ozcicek A, Timuroglu A, Bakirci EM, Hamur H, Ozcicek F, Turkmen K. Association of epicardial adipose tissue, neutrophil-to-lymphocyte ratio and platelet-to-lymphocyte ratio with diabetic nephropathy. Int J Clin Exp Med. 2014 Jul 15;7(7):1794-801. eCollection 2014. PMID 25126182
- [Background] Hozo SP, Djulbegovic B, Hozo I. Estimating the mean and variance from the median, range, and the size of a sample. BMC Med Res Methodol. 2005 Apr 20;5:13. doi: 10.1186/1471-2288-5-13. PMID 15840177
- [Background] HILLER A, GREIF RL, BECKMAN WW. Determination of protein in urine by the biuret method. J Biol Chem. 1948 Dec;176(3):1421-9. No abstract available. PMID 18098591